CLINICAL TRIAL: NCT02747836
Title: Ultrasound Analysis of Human Carpal Tunnel Synovium
Brief Title: Ultrasound Analysis of Human Carpal Tunnel System
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter C. Amadio, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 06-002950
Record Dates: First submitted 2016-04-11; First posted 2016-04-22 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Ultrasound of the wrist
  Interventions: Other: Ultrasound of the wrist
- Participants with Carpal Tunnel Syndrome: Ultrasound of the wrist
  Interventions: Other: Ultrasound of the wrist

INTERVENTIONS:
Other: Ultrasound of the wrist — using sound waves to create images capturing the movement of the SSCT and flexor tendon and transformation of the median nerve in the wrist

SUMMARY:
This study evaluates the ability of ultrasound to measure the movement of tendons and nerves within the human carpal tunnel.

DETAILED DESCRIPTION:
The overall goal of this project is to develop a novel ultrasonographic method to characterize the subsynovial connective tissue (SSCT) and detect differences between SSCT, median nerve and tendon motion for the evaluation and diagnosis of patients suspected of having carpal tunnel syndrome (CTS). CTS is usually diagnosed late in its evolution, by measuring electrophysiological changes in median nerve function. Once these changes have occurred, surgery is often the only effective treatment. At an earlier stage of evolution, non-surgical treatment might be more effective. Although ultrasonography and magnetic resonance imaging (MRI) have recently been used to measure changes in median nerve shape in CTS, such approaches also only capture late changes. Thus, a method for detection of CTS that could identify pathology before function or structure of the nerve is compromised could prevent significant morbidity and transition to a permanent neuropathy. One promising opportunity is presented in the subsynovial connective tissue (SSCT), which surrounds the tendons in the carpal tunnel. One of the most characteristic findings in surgically treated patients with CTS is a non-inflammatory fibrosis of the SSCT. Some investigators have suggested that the SSCT may be the cause of the nerve compression in CTS. In our previous work, the investigators have demonstrated differences in the mechanical properties, motion and thickness of the SSCT in patients with CTS compared to normals. More recently, an animal model has been described in which the structural changes in the SSCT have been shown to precede the changes in nerve function.

The investigators have demonstrated in cadaver studies that the normal SSCT can be imaged by ultrasound, and its motion, velocity, and thickness distinguished from that of the nearby tendon and nerve. Here the investigators propose to leverage this work, and study the ability of ultrasound to detect SSCT thickness and motion in individuals with and without CTS. Based on our preliminary research, the investigators formulate the following central hypothesis: An increase in SSCT thickness and changes in sliding velocities of the SSCT with respect to the corresponding tendon are indicative of CTS. In addition, this material property change at SSCT affects median nerve motions and transformations. This is because the SSCT becomes fibrotic in CTS, and the fibrosis alters the normal SSCT-median nerve-tendon functional relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be selected from among those undergoing diagnostic work up for CTS in the pre-treatment period. CTS diagnosis will be confirmed clinically and by nerve conduction study

Exclusion Criteria:

* The following disorders will be criteria for exclusion:

  * any history of cervical radiculopathy
  * rheumatoid arthritis
  * osteoarthritis
  * degenerative joint disease
  * flexor tendinitis
  * gout hemodialysis
  * sarcoidosis
  * peripheral nerve disease
  * amyloidosis
  * traumatic injuries to the ipsilateral arm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 volunteers without a history of carpal tunnel syndrome and 120 adult patients with carpal tunnel syndrome between the ages of 18 and 85 will be recruited. Patients and volunteers will be age and gender matched
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2008-04-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Study the ability of ultrasound to detect differences in SSCT thickness in individuals with and without CTS. | at the time of study enrollment. patients are enrolled only for the purpose of obtaining a single imaging study.
  Measure and evaluate SSCT thickness

SECONDARY OUTCOMES:
study the ability to detect differences in median nerve and tendon motion in the transverse plane of individuals with and without carpal tunnel syndrome | at time of enrollment. patients are enrolled only for the purpose of obtaining a single imaging study.
  measure displacement of tendons and nerves and the carpal tunnel in the dorsal-palmar and radioulnar directions
Study the ability of ultrasound to detect differences in SSCT motion in individuals with and without CTS. | at the time of study enrollment. patients are enrolled only for the purpose of obtaining a single imaging study.
  Measure and evaluate changes in sliding velocities of the SSCT with respect to the corresponding tendon

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified IPD can be requested from the PI
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at close of study
Access Criteria: upon request

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials